CLINICAL TRIAL: NCT04871737
Title: Dose-escalation, Open-label, Non-randomized Phase I Study to Evaluate the Safety and Immunogenicity of Three Concentrations of a rNDV Vaccine Against SARS-CoV-2 Administered by the Intranasal and Intramuscular Route to Healthy Volunteers
Brief Title: Study of a Live rNDV Based Vaccine Against COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorio Avi-Mex, S.A. de C.V. (Industry)
Collaborators: National Council of Science and Technology, Mexico (Other); Agencia Mexicana de Cooperación Internacional para el Desarrollo. AMEXCID (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: AVX-SARS-CoV-2-VAC-001
Record Dates: First submitted 2021-04-21; First posted 2021-05-04 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: SARS-CoV-2 Infection
Keywords: Newcastle Disease Virus; rNDV; COVID-19; SARS-Cov-2 Vaccine; COVID-19 Vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Patients will be assigned in the order they enter the study into nine treatment groups according to dose and route of administration.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Low Dose, IM-IM (Experimental): Group 1. Dose: 10 7.0-7.49 EID 50/dose. Both first and second administration by the intramuscular route, separated by 21 days.
  Interventions: Biological: Recombinant NDV Vectored Vaccine for SARS-CoV-2
- Intermediate dose, IM-IM (Experimental): Group 2. Dose: 10 7.5-7.99 EID 50/dose. Both first and second administration by the intramuscular route, separated by 21 days
  Interventions: Biological: Recombinant NDV Vectored Vaccine for SARS-CoV-2
- High dose, IM-IM (Experimental): Group 3. Dose: 10 8.0-8.49 EID 50/dose. Both first and second administration by the intramuscular route, separated by 21 days.
  Interventions: Biological: Recombinant NDV Vectored Vaccine for SARS-CoV-2
- Low dose, IN-IN (Experimental): Group 4. Dose: 10 7.0-7.49 EID 50/dose. Both first and second administration by the intranasal route, separated by 21 days
  Interventions: Biological: Recombinant NDV Vectored Vaccine for SARS-CoV-2
- Intermediate dose, IN-IN (Experimental): Group 5. Dose: 10 7.5-7.99 EID 50/dose. Both first and second administration by the intranasal route, separated by 21 days
  Interventions: Biological: Recombinant NDV Vectored Vaccine for SARS-CoV-2
- High dose, IN-IN (Experimental): Group 6. Dose: 10 8.0-8.49 EID 50/dose. Both first and second administration by the intranasal route, separated by 21 days
  Interventions: Biological: Recombinant NDV Vectored Vaccine for SARS-CoV-2
- Low dose, IN-IM (Experimental): Group 7. Dose: 10 7.0-7.49 EID 50/dose. First administration by the intranasal route and second administration by the intramuscular route, separated by 21 days
  Interventions: Biological: Recombinant NDV Vectored Vaccine for SARS-CoV-2
- Intermediate dose, IN-IM (Experimental): Group 8. Dose: 10 7.5-7.99 EID 50/dose. First administration by the intranasal route and second administration by the intramuscular route, separated by 21 days
  Interventions: Biological: Recombinant NDV Vectored Vaccine for SARS-CoV-2
- High dose, IN-IM (Experimental): Group 9. Dose: 10 8.0-8.49 EID 50/dose. First administration by the intranasal route and second administration by the intramuscular route, separated by 21 days
  Interventions: Biological: Recombinant NDV Vectored Vaccine for SARS-CoV-2
- High dose, IM (Experimental): Group 10. Dose: 10 8.0-8.49 EID 50/dose. 3rd administration by the intramuscular route to all the volunteers who agree to participate
  Interventions: Biological: Recombinant NDV Vectored Vaccine for SARS-CoV-2

INTERVENTIONS:
Biological: Recombinant NDV Vectored Vaccine for SARS-CoV-2 — Recombinant Newcastle Disease Virus Vectored Vaccine for SARS-CoV-2

SUMMARY:
This is a Phase 1, open-label, non-randomized, dose-escalation study using three doses and two schemes of administration of a recombinant vaccine against SARS-CoV-2 based on a viral vector (Newcastle Disease virus) in 90 healthy volunteers at a single research site in Mexico City.

DETAILED DESCRIPTION:
The lack of highly effective treatments against COVID-19 and the social and economic impact that the current pandemic has exerted on public health highlights the uncontested importance of developing vaccines that, in addition to their safety and ability to induce a protective response, are logistically suitable for massive administration across a variety of countries and settings.

This is the first clinical study of the development program of a vaccine based on a unique recombinant viral vector technology that has been successful in the design of avian vaccines and that has no contraindication for use in humans.

The recombinant vaccine subject to research in this study is based on an active viral vector of a recombinant Newcastle Disease virus (rNDV) LaSota strain, in which the gene that codes for the S glycoprotein of SARS-CoV-2 has been inserted.

The Newcastle Disease Virus (NDV) is a paramyxovirus responsible for the Newcastle Disease in birds. There are three main families of NDV according to the level of virulence. The one with the lowest virulence is the lentogenic group. One lentogenic viral strain is LaSota (NDV_LS), which is broadly used in the development of avian vaccines. The LaSota strain seems to replicate only at the site of inoculation and, although it does not reach the lymph nodes, it reduces the induction of pro-inflammatory cytokines while boosting a robust protective immune response. Very importantly, this virus cannot insert itself into the human genome.

One of the key factors for an increased virulence in NDV is the activation of the cleavage site that corresponds to the protein F precursor phenotype. In highly virulent strains, the cleavage is performed by ubiquitous intracellular proteins, which leads to a widespread replication in birds.

However, the cleavage site in attenuated or non-virulent strains is activated by a secretory protease which restrains viral replication to mucosal surfaces. This is the same secretory protease which acts in NDV-LS in humans and non-human primates, limiting viral replication to the upper airways.

It is of note that the NDV genome is non-segmented. For this reason, transcription results in a single-stranded RNA which provides the genome with enough stability to avoid reassortment events. These features underpin the antigenic and genetic stability that have contributed to the success of NDV across decades as a vaccine vector.

The recombinant nature of the viral vector is based in the design and synthesis of a gene that codes for the spike protein in SARS-CoV-2. Such design is based in the sequence of the Wuhan-Hu-1 virus (NC_045512.2) and assembled in silico.

Lentogenic strains like LaSota have been used for more than 70 years of vaccination in avian populations and have proven to be safe and with a remarkable naturally attenuated viral activity. In fact, studies have shown that the insertion of foreign genes into the NDV genome leads to a further reduction of pathogenicity in birds. Furthermore, the rNDV is not excreted in feces and therefore not transmitted from bird to bird. Safety tests with avian rNDV vaccines have shown that doses 10 times higher than the dose suggested in this study are not associated with any pathogenicity.

A rNDV vaccine against SARS-CoV and other emerging infections had been proposed. It has been demonstrated that a rNDV vector expressing the S-protein in the SARS-CoV coronavirus is capable of developing protective immunity without safety concerns when administered to African green monkeys by the intranasal route.

It has been reported that rNDV injected by the IV route in non-human primates (Macaca fascicularis) was not associated with any severe disease or abnormalities in hematological or biochemical lab values.

Recently, in the context of the COVID-19 pandemic, a vaccine based on a S-protein expressing viral vector of the Newcastle Disease virus (NDV) has been studied using both a wild type and a pre-fusion membrane-anchored vector format. These studies were performed in mice and hamster models with two administrations of the vaccine. The tested vaccines induced high levels of neutralizing antibodies when administered by the intramuscular route. Notably, these vaccine prototypes protected mice against a mouse-adapted SARS-CoV-2 challenge: neither viral load nor viral antigen were detected in the lungs.

To produce the rNDV, a cell line is transfected by plasmids that express the whole viral genome that contains the gene in question. The clone of the whole NDV genome is transfected with helper plasmids that code for the viral proteins N, P and L under the control of the bacteriophage T7 RNA-polymerase promoter. The chimeric virus is obtained from the culture and propagated in chicken embryo SPF of 10 days of age, until the original vaccine virus is generated.

The vaccine has been formulated for intranasal and intramuscular administration.

In our study, ninety healthy volunteers with no history of COVID-19, vaccination against SARS-CoV-2 or an activity associated with a higher risk of exposure to SARS-CoV-2 will be assigned sequentially into one of nine treatment groups at a single research site in Mexico City.

These treatment groups correspond to three different doses and three different schemes of administration. All these schemes foresee two vaccine administrations separated by 21 days. 3rd administration by the intramuscular route to all the volunteers who agree to participate (see "Arms and Interventions").

Patients will be followed for efficacy and safety measurements. Efficacy will be measured by circulating and neutralizing IgG and IgM antibodies against the S protein of SARS-CoV-2, IgA titers in nasal mucosa and cytokine-mediated T cell responses. Patient safety will be monitored by the collection of information on adverse events and safety laboratory assessments (mainly hematology and blood chemistry).

The first intervention for each treatment group will be administered in a sequential way to eighteen sentinel subjects. Once all sentinel subjects have received the first intervention and the Safety Data Monitoring Board has determined that safety conditions have been met, the study will proceed to enroll the rest of the subjects until a total of 90 participants is reached.

Statistical tests will be applied to each treatment group with similar baseline characteristics. For continuous variables Student's t distribution and ANOVA will be used to compare mean values, while chi-square and Fisher´s exact test will be used to assess categorical values.

There are three working hypotheses to be tested, one for each scheme of administration. They can be consolidated as follows : The recombinant anti-SARS-CoV-2 vaccine based on a viral vector (rNDV) administered [two times by the intramuscular route / two times by the intranasal route / the first by the intranasal route and the second by the intramuscular route] is safe (i.e. an acceptable low profile or reactogenicity: low frequency of mild-to-moderate and no severe local or systemic adverse reactions) and induces a humoral and cellular immune response against SARS-CoV-2 similar (or greater) to that measured in sera from naturally-acquired COVID-19 convalescent individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women ≥18 year-old and ≤55-year-old.
* Signed informed consent.
* No respiratory disease within last 21 days prior to first dose administration.
* Body Mass Index from 18.0 to 29.0 kg/m2.
* Negative RT-PCR for SARS-Cov-2 infection.
* Negative test for anti-SARS-CoV-2 IgM and IgG antibodies.
* O2 saturation ≥92% by pulse oximetry.
* Normal CT scan of thorax.
* No symptoms from clinical history and normal physical exam at screening visit.
* Lab test values within normal ranges for all the following:

Urinalysis. Liver enzymes. Renal function tests. Cholesterol and Triglycerides. Fasting glucose. Hematology.

* Negative test for HBsAg, anti-HCV and anti-HIV antibodies. Negative VDRL test.
* Normal electrocardiogram.
* Negative pregnancy test for women with childbearing potential.
* Agreement of all sexually- active volunteers to use highly effective contraceptives over the study period and up to 30 days after the last administration of the experimental vaccine.
* Commitment from all participants to keep social distancing, use of mask and frequent hand washing with soap or antibacterial gel during the study period.

Exclusion Criteria:

* History of hypersensitivity or allergy to any ingredient of the vaccine.
* History of severe anaphylactic reaction.
* History of seizures.
* History of chronic diseases or cancer.
* Vaccination against SARS-CoV-2 with approved or experimental vaccines.
* Participation in any other study with an experimental intervention within the last 3 months.
* Administration of any other drug or herbal preparation within the last 30 days.
* Any vaccine administered within the last 30 days, including influenza vaccine.
* Fever at the time of entry.
* Blood transfusion or blood components transfusion within the last 4 months.
* Regular activity related to work, social interaction or entertainment that represents an exposure to SARS-Cov-2 higher than that of the general population, as per investigator judgement.
* Drug and alcohol abuse.
* Any medical or not medical condition that could interfere with patient safety, study compliance or data interpretation, as per investigator judgement.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-08-21 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Safety: adverse events | Day 2
  Incidence of adverse events
Safety: adverse events | Day 3
  Incidence of adverse events
Safety: adverse events | Day 4
  Incidence of adverse events
Safety: adverse events | Day 5
  Incidence of adverse events
Safety: adverse events | Day 6
  Incidence of adverse events
Safety: adverse events | Day 7
  Incidence of adverse events
Safety: adverse events | Day 14
  Incidence of adverse events
Safety: adverse events | Day 21
  Incidence of adverse events
Safety: adverse events | Day 28
  Incidence of adverse events
Safety: adverse events | Day 35
  Incidence of adverse events
Safety: adverse events | Day 42
  Incidence of adverse events
Safety: adverse events | Day 90
  Incidence of adverse events
Safety: adverse events | Day 180
  Incidence of adverse events
Safety: adverse events | Day 365
  Incidence of adverse events
Safety: Pregnancy test | Day 1
  Blood hCG (mUI/mL)
Safety: Pregnancy test | Day 14
  Blood hCG
Safety: Urinalysis | Day 14
  Qualitative and by sediment examination
Safety: Oxygen saturation | Day 14
  Pulse oximetry (%)

SECONDARY OUTCOMES:
Titers of circulating anti-SARS-CoV2 antibodies | Day 14
  Serum IgG, IgM
Titers of circulating anti-SARS-CoV2 antibodies | Day 21
  Serum IgG, IgM
Titers of circulating anti-SARS-CoV2 antibodies | Day 28
  Serum IgG, IgM
Titers of circulating anti-SARS-CoV2 antibodies | Day 35
  Serum IgG, IgM
Titers of circulating anti-SARS-CoV2 antibodies | Day 42
  Serum IgG, IgM
Titers of circulating anti-SARS-CoV2 antibodies | Day 90
  Serum IgG, IgM
Titers of circulating anti-SARS-CoV2 antibodies | Day 180
  Serum IgG, IgM
Titers of neutralizing anti-SARS-Cov-2 antibodies | Day 14
  Serum IgG, IgM
Titers of neutralizing anti-SARS-Cov-2 antibodies | Day 21
  Serum IgG, IgM
Titers of neutralizing anti-SARS-Cov-2 antibodies | Day 28
  Serum IgG, IgM
Titers of neutralizing anti-SARS-Cov-2 antibodies | Day 42
  Serum IgG, IgM
Titers of neutralizing anti-SARS-Cov-2 antibodies | Day 90
  Serum IgG, IgM
Titers of neutralizing anti-SARS-Cov-2 antibodies | Day 180
  Serum IgG, IgM
Titers of neutralizing anti-SARS-Cov-2 antibodies | Day 365
  Serum IgG, IgM
Titers of mucosal IgA | Day 14
  Mucosal IgA
Titers of mucosal IgA | Day 21
  Mucosal IgA
Titers of mucosal IgA | Day 28
  Mucosal IgA
Titers of mucosal IgA | Day 42
  Mucosal IgA
Titers of mucosal IgA | Day 90
  Mucosal IgA
Titers of mucosal IgA | Day 180
  Mucosal IgA
Titers of mucosal IgA | Day 365
  Mucosal IgA
T-cell elicited responses | Day 14
  Percentage of cells expressing IL2, TNFalpha and IFNgamma by flow cytometry after challenge with spike protein
T-cell elicited responses | Day 21
  Percentage of cells expressing IL2, TNFalpha and IFNgamma by flow cytometry after challenge with spike protein
T-cell elicited responses | Day 28
  Percentage of cells expressing IL2, TNFalpha and IFNgamma by flow cytometry after challenge with spike protein
T-cell elicited responses | Day 42
  Percentage of cells expressing IL2, TNFalpha and IFNgamma by flow cytometry after challenge with spike protein
T-cell elicited responses | Day 90
  Percentage of cells expressing IL2, TNFalpha and IFNgamma by flow cytometry after challenge with spike protein
T-cell elicited responses | Day 180
  Percentage of cells expressing IL2, TNFalpha and IFNgamma by flow cytometry after challenge with spike protein
T-cell elicited responses | Day 365
  Percentage of cells expressing IL2, TNFalpha and IFNgamma by flow cytometry after challenge with spike protein
Titers of circulating anti-SARS-CoV2 antibodies | Day 14 after application
  Serum IgG, IgM after 3rd dose
Titers of circulating anti-SARS-CoV2 antibodies | Day 42 after application
  Serum IgG, IgM after 3rd dose
Titers of circulating anti-SARS-CoV2 antibodies | Day 90 after application
  Serum IgG, IgM after 3rd dose
Titers of neutralizing anti-SARS-Cov-2 antibodies | Day 14 after application
  Serum IgG, IgM after 3rd dose
Titers of neutralizing anti-SARS-Cov-2 antibodies | Day 42 after application
  Serum IgG, IgM after 3rd dose
Titers of neutralizing anti-SARS-Cov-2 antibodies | Day 90 after application
  Serum IgG, IgM after 3rd dose
Titers of secretory IgA | Day 14 after application
  Mucosal IgA after 3rd dose
Titers of secretory IgA | Day 42 after application
  Mucosal IgA after 3rd dose

OTHER OUTCOMES:
Safety: adverse events [Exploratory Outcomes] | 365 + 14 days after application
  Incidence of adverse events after 3rd dose
Safety: adverse events [Exploratory Outcomes] | 365 + 42 days after application
  Incidence of adverse events after 3rd dose
Safety: adverse events [Exploratory Outcomes] | 365 + 90 days after application
  Incidence of adverse events after 3rd dose

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Ponce de Leon, MD, Principal Investigator — Universidad Nacional Autonoma de Mexico
Locations (1):
- Hospital Medica Sur, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Honda K, Sakaguchi S, Nakajima C, Watanabe A, Yanai H, Matsumoto M, Ohteki T, Kaisho T, Takaoka A, Akira S, Seya T, Taniguchi T. Selective contribution of IFN-alpha/beta signaling to the maturation of dendritic cells induced by double-stranded RNA or viral infection. Proc Natl Acad Sci U S A. 2003 Sep 16;100(19):10872-7. doi: 10.1073/pnas.1934678100. Epub 2003 Sep 5. PMID 12960379
- [Background] Czegledi A, Ujvari D, Somogyi E, Wehmann E, Werner O, Lomniczi B. Third genome size category of avian paramyxovirus serotype 1 (Newcastle disease virus) and evolutionary implications. Virus Res. 2006 Sep;120(1-2):36-48. doi: 10.1016/j.virusres.2005.11.009. PMID 16766077
- [Background] DiNapoli JM, Kotelkin A, Yang L, Elankumaran S, Murphy BR, Samal SK, Collins PL, Bukreyev A. Newcastle disease virus, a host range-restricted virus, as a vaccine vector for intranasal immunization against emerging pathogens. Proc Natl Acad Sci U S A. 2007 Jun 5;104(23):9788-93. doi: 10.1073/pnas.0703584104. Epub 2007 May 29. PMID 17535926
- [Background] Buijs PR, van Amerongen G, van Nieuwkoop S, Bestebroer TM, van Run PR, Kuiken T, Fouchier RA, van Eijck CH, van den Hoogen BG. Intravenously injected Newcastle disease virus in non-human primates is safe to use for oncolytic virotherapy. Cancer Gene Ther. 2014 Nov;21(11):463-71. doi: 10.1038/cgt.2014.51. Epub 2014 Sep 26. PMID 25257305
- [Background] Sun W, Leist SR, McCroskery S, Liu Y, Slamanig S, Oliva J, Amanat F, Schafer A, Dinnon KH 3rd, Garcia-Sastre A, Krammer F, Baric RS, Palese P. Newcastle disease virus (NDV) expressing the spike protein of SARS-CoV-2 as a live virus vaccine candidate. EBioMedicine. 2020 Dec;62:103132. doi: 10.1016/j.ebiom.2020.103132. Epub 2020 Nov 21. PMID 33232870
- [Background] Sun W, McCroskery S, Liu WC, Leist SR, Liu Y, Albrecht RA, Slamanig S, Oliva J, Amanat F, Schafer A, Dinnon KH 3rd, Innis BL, Garcia-Sastre A, Krammer F, Baric RS, Palese P. A Newcastle Disease Virus (NDV) Expressing a Membrane-Anchored Spike as a Cost-Effective Inactivated SARS-CoV-2 Vaccine. Vaccines (Basel). 2020 Dec 17;8(4):771. doi: 10.3390/vaccines8040771. PMID 33348607
- [Derived] Ponce-de-Leon S, Torres M, Soto-Ramirez LE, Calva JJ, Santillan-Doherty P, Carranza-Salazar DE, Carreno JM, Carranza C, Juarez E, Carreto-Binaghi LE, Ramirez-Martinez L, Paz De la Rosa G, Vigueras-Moreno R, Ortiz-Stern A, Lopez-Vidal Y, Macias AE, Torres-Flores J, Rojas-Martinez O, Suarez-Martinez A, Peralta-Sanchez G, Kawabata H, Gonzalez-Dominguez I, Martinez-Guevara JL, Sun W, Sarfati-Mizrahi D, Soto-Priante E, Chagoya-Cortes HE, Lopez-Macias C, Castro-Peralta F, Palese P, Garcia-Sastre A, Krammer F, Lozano-Dubernard B. Interim safety and immunogenicity results from an NDV-based COVID-19 vaccine phase I trial in Mexico. NPJ Vaccines. 2023 May 10;8(1):67. doi: 10.1038/s41541-023-00662-6. PMID 37164959
- [Derived] Ponce-de-Leon S, Torres M, Soto-Ramirez LE, Calva JJ, Santillan-Doherty P, Carranza-Salazar DE, Carreno JM, Carranza C, Juarez E, Carreto-Binaghi LE, Ramirez-Martinez L, Paz-De la Rosa G, Vigueras-Moreno R, Ortiz-Stern A, Lopez-Vidal Y, Macias AE, Torres-Flores J, Rojas-Martinez O, Suarez-Martinez A, Peralta-Sanchez G, Kawabata H, Gonzalez-Dominguez I, Martinez-Guevara JL, Sun W, Sarfati-Mizrahi D, Soto-Priante E, Chagoya-Cortes HE, Lopez-Macias C, Castro-Peralta F, Palese P, Garcia-Sastre A, Krammer F, Lozano-Dubernard B. Safety and immunogenicity of a live recombinant Newcastle disease virus-based COVID-19 vaccine (Patria) administered via the intramuscular or intranasal route: Interim results of a non-randomized open label phase I trial in Mexico. medRxiv [Preprint]. 2022 Feb 9:2022.02.08.22270676. doi: 10.1101/2022.02.08.22270676. PMID 35169806